CLINICAL TRIAL: NCT01796938
Title: Open, Non-randomized, Sequential Group Comparison to Investigate the Pharmacokinetics, Safety, and Tolerability of 100 mg SPM 927 in Male and Female Subjects With Renal Impairment Including Subjects Requiring Dialysis Compared With Male and Female Healthy Subjects Following Single-dose Administration
Brief Title: Study to Evaluate the Pharmacokinetics, Safety, Tolerability of Single Dose Lacosamide in Subjects With Renal Impairment Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: SP0641
Record Dates: First submitted 2013-02-19; First posted 2013-02-22 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2013-02

CONDITIONS: Healthy; Renal Impairment
Keywords: Lacosamide; Vimpat; Single Dose; Pharmacokinetics; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1: Healthy subjects (Experimental): Single dose of 100 mg Lacosamide
  Interventions: Drug: Lacosamide tablet
- Group 2: Subjects with mild renal insufficiency (Experimental): Single dose of 100 mg Lacosamide
  Interventions: Drug: Lacosamide tablet
- Group 3: Subjects with moderate renal insufficiency (Experimental): Single dose of 100 mg Lacosamide
  Interventions: Drug: Lacosamide tablet
- Group 4: Subjects with severe renal insufficiency (Experimental): Single dose of 100 mg Lacosamide
  Interventions: Drug: Lacosamide tablet
- Group 5: Subjects with end stage renal insufficiency (Experimental): Single dose of 100 mg Lacosamide
  Interventions: Drug: Lacosamide tablet

INTERVENTIONS:
Drug: Lacosamide tablet — Single dose of 100 mg Lacosamide tablet
  Other Names: Vimpat

SUMMARY:
To investigate the Pharmacokinetics (PK) of oral administered Lacosamide in renal impaired subjects and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject was informed and given ample time and opportunity to think about his/her participation and had given his/her written informed consent
* Subject was willing and able to comply with all trial requirements
* Subject was a male or female Caucasian, between 18 and 70 years of age (inclusive)
* If female, subject was of non-childbearing potential (post-menopausal or hysterectomized) or was using medically adequate contraception
* If female of childbearing potential, subject had a negative pregnancy test
* Subject had a Body Mass Index (BMI) between 20 and 34 kg/m2 (inclusive)
* Subject was healthy without clinically relevant cardiovascular, renal, gastrointestinal, hepatic, metabolic, endocrine, neurological, or psychiatric abnormalities detected during Eligibility Assessment (EA)

Subjects with renal impairment also had to fulfill the following inclusion criteria:

* Subject had no clinically relevant cardiovascular or endocrine findings during EA
* Subject had a renal impairment. The subjects were assigned to 1 of the following treatment groups according to Creatinine Clearance (CLCr) values determined 2 to 7 days prior to dosing:
* Group 2: 80 mL/min > CLCr ≥ 50 mL/min (subjects with mild renal impairment)
* Group 3: 50 mL/min > CLCr ≥ 30 mL/min (subjects with moderate renal impairment)
* Group 4: CLCr < 30 mL/min (subjects with severe renal impairment, not on dialysis between 2 weeks before EA and end of the trial)

Inclusion criteria for Group 5:

* Subject was informed and given ample time and opportunity to think about his/her participation and had given his/her written informed consent
* Subject was willing and able to comply with all trial requirements
* Subject was a male or female Caucasian, between 18 and 70 years of age (inclusive)
* If female, subject was of non-childbearing potential (post-menopausal or hysterectomized) or was using medically adequate contraception
* If female of childbearing potential, subject had a negative pregnancy test
* Subject had a BMI between 20 and 34 kg/m2 (inclusive)
* Subject had no clinically relevant cardiovascular or endocrine findings during EA
* Subject had an endstage renal disease (CLCr < 15 mL/min, determined approximately 2 to 7 days before first dosing) treated with extracorporal hemodialysis for at least 4 months

Exclusion Criteria:

Healthy subjects:

* Subject had previously participated in this trial
* Subject had participated in another trial of an investigational product within the last 3 months or was currently participating in another trial of an investigational product
* Subject had donated blood or had a comparable blood loss (> 500 mL) within the last 3 months prior to EA
* Subject smoked more than 5 cigarettes per day or had done so within the 6 months prior to commencement of this trial
* Subject had a history of chronic alcohol or drug abuse within the last 6 months prior to commencement of this trial
* Subject consumed more than 40 g of alcohol/day (amount corresponds to 1 L beer/day or 0.5 L wine/day or 120 mL liquor/day)
* Subject had positive tests for alcohol (urine or breath test) or drugs (urine test)
* Subject had clinically relevant changes in the electrocardiogram (ECG), such as second- or third-degree atrioventricular (AV) block, prolongation of the QRS complex over 120 ms or of the corrected QT (QTc) interval > 430 ms (male subjects) or > 450 ms (female subjects)
* Subject had a history or present condition of clinically relevant respiratory or cardiovascular disorders, eg, cardiac insufficiency, coronary heart disease, hypertension, arrhythmia, tachyarrhythmia, or status after myocardial infarction
* Subject had a history or present condition of psychic abnormality, psychiatric or neurologic illness, or autonomic neuropathy that, in the opinion of the Investigator, could have jeopardized or would have compromised the subject's ability to participate in the trial
* Subject had a history or present condition of seizure disorder
* Subject had a history or present condition of malignancy
* Subject had a history or present condition of renal disorders (albuminuria, chronic infections) or renal impairment
* Subject had a history or present condition of Diabetes Mellitus or thyroid dysfunction, especially Hyperthyreosis, or other endocrine disorders
* Subject had a clinically relevant allergy
* Subject had a known or suspected drug hypersensitivity, in particular to the trial medication
* Subject was taking any concomitant medication currently or within 2 weeks prior to the first day of dosing (with the exception of oral contraceptives and Paracetamol [maximum allowed dose: 1000 mg/dose], which were allowed up to 48 hours prior to dosing); further exceptions could be made if the Investigator and the sponsor jointly considered the medication as acceptable
* Subject was tested positive for human immunodeficiency virus 1/2 antibodies (HIV-1/2-Ab), hepatitis B surface antigen (HBs-Ag), or hepatitis C virus antibody (HCV-Ab)
* Subject had any clinically relevant abnormality in the physical examination or in vital sign measurements (systolic blood pressure > 150 mmHg or < 100 mmHg, diastolic blood pressure > 95 mmHg or < 60 mmHg, pulse rate > 100 beats per minute (bpm) or < 50 bpm)
* Subject had a clinically relevant deviation from the norm in the clinical chemistry, hematology, or urinalysis evaluations

Exclusion criteria for Groups 2-4:

* Exclusion criteria 1 to 12 for healthy subjects also applied to subjects with renal impairment
* Subject had a clinically relevant allergy
* Subject had a known or suspected drug hypersensitivity, in particular to the trial medication
* Subject was taking any concomitant medication currently or within 2 weeks prior to dosing that could have interfered with the investigational product
* Subject was tested positive for HIV-1/2-Ab, HBs-Ag, or HCV-Ab
* Subject had any clinically relevant abnormality in the physical examination or in vital sign measurements (systolic blood pressure > 180 mmHg or < 100 mmHg, diastolic blood pressure > 110 mmHg, pulse rate > 100 bpm or < 60 bpm)
* Subject had a clinically relevant deviation from the norm in the clinical chemistry, hematology or urinalysis evaluations other than expected for a subject with renal impairment, eg, hemoglobin < 8.0 g/dL

Exclusion criteria for Group 5:

* Exclusion criteria 1 to 12 for healthy subjects also applied to subjects in Group 5
* Subject had a clinically relevant allergy
* Subject had a known or suspected drug hypersensitivity, in particular to the trial medication
* Subject was tested positive for HIV-1/2-Ab, HBs-Ag, or HCV-Ab
* Subject was taking any concomitant medication that might interfere with the investigational product currently or within 2 weeks prior to dosing
* Subject had any clinically relevant abnormality in the physical examination or in vital sign measurements (systolic blood pressure > 200 mmHg [predialysis value] or < 100 mmHg, diastolic blood pressure > 110 mmHg, pulse rate > 100 bpm or < 60 bpm)
* Subject had a clinically relevant deviation from the norm in the clinical chemistry, hematology, or urinalysis evaluations other than expected for a patient with renal impairment, eg, hemoglobin < 8.0 g/dL

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-06; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Area under the Lacosamide plasma concentration time curve from 0 to the last quantifiable data point (AUC(0-tz)) | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5
Measured maximal concentration (Cmax) of Lacosamide | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5
Area under the Lacosamide plasma concentration-time curve from 0 to the last quantifiable data point (AUC (0-tz)), normalized by body weight | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5
Measured maximal concentration (Cmax, norm) of Lacosamide normalized by body weight | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5

SECONDARY OUTCOMES:
Time of observed maximum (tmax) of Lacosamide concentration | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5
Time of observed maximum (tmax) of Lacosamide metabolite (SPM12809) concentration | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5
Terminal half-life (t1/2) of Lacosamide | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5
Terminal half-life (t1/2) of Lacosamide metabolite (SPM12809) | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5
Apparent total clearance (CL/f) of Lacosamide from plasma | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5
Area under the lacosamide metabolite (SPM12809) plasma concentration-time curve from 0 to the last quantifiable data point (AUC(0-tz)) | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5
Amount of Lacosamide excreted in urine from 0 to defined time point (Ae(0-48)) (t=48 hours) | Day 1 to Day 3 of study
  Urine sampling predose, 0-4, 4-8, 8-12, 12-24, 24-36, and 36-48 hours postdose
Amount of Lacosamide metabolite (SPM12809) excreted in urine from 0 to defined time point (Ae(0-48)) (t=48 hours) | Day 1 to Day 3 of study
  Urine sampling predose, 0-4, 4-8, 8-12, 12-24, 24-36, and 36-48 hours postdose
Measured maximal concentration (Cmax) of Lacosamide metabolite (SPM12809) | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5
Area under the Lacosamide metabolite (SPM12809) plasma concentration time curve from 0 to the last quantifiable data point (AUC(0-tz)), normalized by body weight | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5
Measured maximal Lacosamide metabolite (SPM12809) concentration (Cmax,norm), normalized by body weight | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5
Terminal half-life (t1/2) of Lacosamide in urine | Day 1 to Day 3 of study
  Urine sampling predose, 0-4, 4-8, 8-12, 12-24, 24-36, and 36-48 hours postdose
Lacosamide concentration in dialysis inlet line (Cin) | From 4 hours up to 6 hours postdose
  Dialysis samples collected 4 hours and 6 hours after administration (1.5 hours and 3.5 hours after start of dialysis)
Lacosamide metabolite (SPM12809) concentration in dialysis inlet line (Cin) | From 4 hours up to 6 hours postdose
  Dialysis samples collected 4 hours and 6 hours after administration (1.5 hours and 3.5 hours after start of dialysis)
Lacosamide concentration in dialysis outlet line (Cout) | From 4 hours up to 6 hours postdose
  Dialysis samples collected 4 hours and 6 hours after administration (1.5 hours and 3.5 hours after start of dialysis)
Lacosamide metabolite (SPM12809) concentration in dialysis outlet line (Cout) | From 4 hours up to 6 hours postdose
  Dialysis samples collected 4 hours and 6 hours after administration (1.5 hours and 3.5 hours after start of dialysis)
Extraction rate (E) of Lacosamide | From 4 hours up to 6 hours postdose
  Dialysis samples collected 4 hours and 6 hours after administration (1.5 hours and 3.5 hours after start of dialysis)
Extraction rate (E) of Lacosamide metabolite (SPM12809) | From 4 hours up to 6 hours postdose
  Dialysis samples collected 4 hours and 6 hours after administration (1.5 hours and 3.5 hours after start of dialysis)
Dialysis clearance (CLdial) of Lacosamide | From 4 hours up to 6 hours postdose
  Dialysis samples collected 4 hours and 6 hours after administration (1.5 hours and 3.5 hours after start of dialysis)
Dialysis clearance (CLdial) of Lacosamide metabolite (SPM12809) | From 4 hours up to 6 hours postdose
  Dialysis samples collected 4 hours and 6 hours after administration (1.5 hours and 3.5 hours after start of dialysis)
Rate constant of Lacosamide elimination | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5
Rate constant of Lacosamide metabolite (SPM12809) elimination | Day 1 to Day 5 of study
  Blood sampling at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after single dose administration; > 24 hours excluded for group 5

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (2):
- Germany (2):
  - 1, Cologne
  - 2, Rendsburg

REFERENCES:
- [Derived] Cawello W, Fuhr U, Hering U, Maatouk H, Halabi A. Impact of impaired renal function on the pharmacokinetics of the antiepileptic drug lacosamide. Clin Pharmacokinet. 2013 Oct;52(10):897-906. doi: 10.1007/s40262-013-0080-7. PMID 23737404